CLINICAL TRIAL: NCT06608108
Title: The Clinical Efficacy of CT-Guided All-in-One Adaptive Emergency Radiotherapy for Spinal Cord Compression Caused by Spinal Metastases
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 551-02
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-10

CONDITIONS: Malignant Spinal Cord Compression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Non-interventional studies
  Interventions: Other: Non-intervention

INTERVENTIONS:
Other: Non-intervention — Non-intervention

SUMMARY:
The aim of this study is to implement a new protocol for concurrent and sequential dose-escalation radiotherapy based on CT-guided all-in-one adaptive emergency radiotherapy for spinal cord compression due to spinal metastases (MSCC). This protocol is designed to assess the clinical efficacy in MSCC patients, with the goals of improving local control rates, functional relief, and optimizing treatment outcomes and safety. The study also seeks to provide reliable data and guidance for future radiotherapy protocol design and clinical practice. Additionally, the study records and analyzes the treatment time required for the all-in-one emergency radiotherapy, aiding in the evaluation of its operational efficiency and clinical feasibility, and providing data support for its broader adoption and dissemination.

DETAILED DESCRIPTION:
Spinal Cord Compression Syndrome (SCCS) is a clinical syndrome caused by space-occupying lesions within the spine or spinal canal. These lesions exert pressure on the spinal cord, spinal nerve roots, and the blood vessels supplying the spinal cord, leading to neurological deficits and, ultimately, spinal cord dysfunction. Spinal cord compression caused by primary malignant tumors or distant metastases of malignant tumors is referred to as Malignant Spinal Cord Compression (MSCC), a common complication in advanced cancer. Approximately 40% of cancer patients develop metastatic spinal disease, and 10-20% of these patients will experience spinal cord compression symptoms. MSCC is characterized by its rapid onset, short course, and fast progression. Early symptoms often manifest as localized or radiating pain. As the condition progresses, patients may experience muscle weakness, sensory deficits, impaired voluntary movement (particularly loss of bowel and bladder control), and even complete paralysis. If not diagnosed and treated promptly, MSCC can severely affect quality of life of patients.

Radiation therapy is one of the most commonly used and effective treatments for MSCC. Radiotherapy reduces tumor burden, alleviates localized bone pain, prevents pathological fractures and vertebral collapse, promotes the healing of pathological fractures, and relieves spinal cord compression, thereby improving mobility, function, and quality of life of patients. However, conventional radiotherapy workflows are complex and involve multiple steps. Patients typically need to visit different departments multiple times and may face days of waiting before receiving treatment, which is far from ideal in the emergency context of MSCC. The domestic innovative radiotherapy equipment, uRT-linac506C, was developed to address this need. It integrates diagnostic-grade spiral CT and linear accelerator technology into a single workflow, allowing for seamless, rapid transitions from simulation, CT scanning, intelligent contouring and modification of tumor targets and organs-at-risk, to treatment plan design, evaluation, verification, and implementation of the first radiation therapy. Without compromising standardized procedures, this significantly shortens waiting and treatment times, realizing All-in-One image-guided, diagnosis-treatment integration that seamlessly connects the various stages of radiotherapy. This approach reduces the time from patient positioning to treatment from several days with conventional radiotherapy to approximately 30 minutes, enabling rapid and precise radiation therapy to relieve spinal cord compression and improve patient outcomes. Investigators refer to this integrated approach as All-in-One emergency radiotherapy.

Although radiotherapy has become the primary treatment for spinal cord compression (especially when surgery is not feasible), emergency radiotherapy has significantly improved the timeliness and effectiveness of treatment, allowing patients to receive rapid relief and care in urgent situations and preventing severe consequences from delayed treatment. However, there is still debate about the specific implementation of radiation therapy for spinal metastases. Various fractionation regimens have been reported in the literature, ranging from single-fraction to multi-fraction radiation therapy. There is no consensus on the optimal treatment regimen for bone metastases in terms of treatment volume, total dose, or fractionation. For patients with a short expected survival, shorter courses of radiotherapy (1-5 fractions, with doses ranging from 8 to 20 Gy) are commonly used to reduce treatment time and minimize patient suffering. For patients with a longer expected survival (e.g., more than 6 months), the risk of disease progression or in-field recurrence must be considered, and longer courses of radiotherapy, such as the commonly used 10 × 3 Gy regimen, are more appropriate.

In previous large retrospective studies, patient survival was not considered, and many patients did not live long enough to experience local recurrence, which may have led to biased results in local control. Therefore, it is reasonable to investigate whether patients with a longer prognosis can benefit from increased radiation doses (beyond the traditional 10 × 3 Gy). For these longer-surviving patients, exploring more precise and individualized radiotherapy regimens is necessary. This may include higher radiation doses and longer treatment durations to achieve better disease control and prolong progression-free and overall survival.

With advances in imaging and radiotherapy technology, Simultaneous Integrated Boost Intensity-Modulated Radiotherapy (SIB-IMRT) has emerged as a radiotherapy technique that applies differential doses to high-risk and low-risk regions within the same radiation field, maximizing normal tissue protection while increasing the dose to the target area. Sequential Boost Radiotherapy involves delivering additional doses to tumors or high-risk areas after the standard radiotherapy course is completed, further increasing the cumulative radiation dose. Based on long-term experience, investigators have developed the ability to escalate the planned gross tumor volume (PGTV) from the traditional 3 Gy per fraction to 4 Gy per fraction while maintaining organ-at-risk dose limits within tolerance. Moreover, the number of sequential boost sessions has been increased from the traditional 10 to 12 sessions, with promising initial results.

Therefore, this study aims to evaluate the efficacy of Simultaneous Integrated and Sequential Boost Radiotherapy in patients with MSCC receiving All-in-One adaptive emergency radiotherapy guided by CT for spinal metastases. Investigators seek to validate its safety and efficacy while also recording and analyzing the overall treatment duration of All-in-One emergency radiotherapy. Ultimately, investigators hope to improve patient quality of life and extend survival, providing scientific evidence and guidance for clinical practice.

Supplement

Dear Professor,

Investigators sincerely appreciate the review of this clinical trial application by the professor. Further clarification regarding the study design and type is provided. Since 2018, the radiation oncology center has employed this dose-fractionation regimen to treat patients with malignant spinal cord compression. Recently, due to clinical demand, an advanced accelerator system integrated with diagnostic-grade CT has been introduced, which is now routinely applied in clinical practice. This study is conducted within this clinical context. All enrolled participants, regardless of their involvement in the study, will receive the same treatment methods and protocols, and the research itself will not influence the treatment. Therefore, this study qualifies as a prospective, non-interventional study.

Should the professor have any further questions or suggestions, please feel free to reach out!

Best regards.

ELIGIBILITY:
Inclusion Criteria:

* (1)Diagnosed with MSCC due to spinal metastases confirmed by imaging (MRI or CT).

  (2)Acute or subacute onset of MSCC. (3)Modified Tokuhashi score for spinal metastases ≥ 9, indicating an expected survival time > 6 months.

  (4)Spinal instability neoplastic score (SINS) ≤ 7, indicating spinal stability. (5)General performance status (Karnofsky score) ≥ 60. (6)No prior radiotherapy or surgical treatment for the spinal metastases before enrollment.

  (7)Patient refuses or is intolerant to surgery. (8)No other severe comorbidities, such as uncontrolled infections or serious cardiopulmonary diseases, that may affect radiotherapy outcomes or increase treatment risks.

  (9)No other active malignancies (except for the primary tumor and spinal metastases) to ensure the study's focus.

  (10)Age 18 years or older. (11)Informed consent obtained from the patient. (12) Accept CT guided spinal cord compression all in one adaptive emergency radiotherapy for spinal metastases.

Exclusion Criteria:

- (1)History of radiotherapy or surgery in the affected spinal region leading to MSCC.

(2)Intolerance to radiotherapy. (3)Severe psychiatric or neurological disorders. (4)Pregnant or breastfeeding women. (5)Clear indications that the affected spinal cord region requires decompression surgery first.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the inclusion and exclusion criteria, 50 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate | The time frame extends from the initiation of radiotherapy until the first recorded local recurrence, with an initial assessment period of 24 months.
  The time frame extends from the initiation of radiotherapy until the first recorded local recurrence, with an initial assessment period of 24 months. Patients will be followed up one month and three months after treatment, and subsequently every three months.

SECONDARY OUTCOMES:
Neurological function assessment | An assessment will be conducted after each radiotherapy session. Patients will be followed up one month and three months after treatment, and subsequently every three months. The initial time frame is 24 months.
  An assessment will be conducted after each radiotherapy session. Patients will be followed up one month and three months after treatment, and subsequently every three months. The initial time frame is 24 months.
Pain evaluation | An assessment will be conducted after each radiotherapy session. Patients will be followed up one month and three months after treatment, and subsequently every three months. The initial time frame is 24 months.
  An assessment will be conducted after each radiotherapy session. Patients will be followed up one month and three months after treatment, and subsequently every three months. The initial time frame is 24 months.
Emergency radiotherapy treatment time | 1 day (Record the duration of each emergency radiotherapy session. The time frame is the period during which the All-in-One emergency radiotherapy is administered.)
  Record the duration of each emergency radiotherapy session. The time frame refers to the period during which All-in-One adaptive emergency radiotherapy is performed, starting from the moment the patient lies on the treatment couch of the linear accelerator for CT localization until the patient completes the treatment and leaves the treatment couch

IPD SHARING:
Plan to Share IPD: No